CLINICAL TRIAL: NCT03414125
Title: Comparing the Effect of a Mailed Outreach Intervention Offering Choice of Colonoscopy or FIT vs. Mailed FIT Alone on Colorectal Cancer Screening Outcomes: A Pragmatic Randomized Control Trial in a Safety Net Health System
Brief Title: Effect of Mailed Invites of Choice of Colonoscopy or FIT vs. Mailed FIT Alone on Colorectal Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Cancer Prevention Research Institute of Texas (Other); Parkland Health and Hospital System (Other)
Responsible Party: Principal Investigator, Amit Singal, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: STU 082016-060; 21985 (Other: UTSouthwestern - Velos); PP160075 (Other Grant/Funding Number: Cancer Prevention and Research Institute of Texas)
Record Dates: First submitted 2018-01-22; First posted 2018-01-29 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; Colon Cancer; FIT Screening Strategy; Colon Screening Strategy; Colorectal Neoplasms; Mass Screening; Health Services Research; Comparative Effectiveness Research
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: Evaluate effect of offering choice of FIT or colonoscopy (n=2,000) compared to FIT alone (n=8,000) on one-time CRC screening completion, repeat screening, and follow-up of abnormal FIT results.
Who Masked: Outcomes Assessor
Masking Description: Single Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FIT Screening Strategy (Active Comparator): Mailed outreach invitation to complete FIT. FIT Strategy invitation includes: 1) invitation letter, 2) test kit (1-sample FIT, simplified instructions on how to perform the test and return mailer with prepaid postage).
  Up to three "live" phone reminders from project staff 2 to 3 weeks after the invitation to encourage screening completion.
  Centralized processes to promote guideline-based follow-up.
  Interventions: Other: FIT Screening Strategy
- Choice Screening Strategy (Experimental): Mailed outreach invitation offering patients the choice to complete either a FIT or schedule a colonoscopy.
  Letter will discuss advantages and disadvantages of FIT vs. colonoscopy but will not recommend a particular test, allowing patients to choose a screening option based on their own preferences.
  Choice Strategy outreach invitation includes: 1) invitation letter, 2) option grid comparing FIT and colonoscopy 3) telephone number for scheduling colonoscopy, and 4) test kit (1-sample FIT, simplified instructions on how to perform the test and return mailer with prepaid postage).
  Up to three "live" phone call reminders from project staff 2 to 3 weeks after the mailed invitation to encourage screening completion.
  Centralized processes to promote guideline-based follow-up.
  Interventions: Other: Choice Screening Strategy

INTERVENTIONS:
Other: FIT Screening Strategy — Mailed outreach invitation to complete FIT. FIT Strategy invitation includes: 1) invitation letter, 2) test kit (1-sample FIT, simplified instructions on how to perform the test and return mailer with prepaid postage).
  Up to three "live" phone reminders from project staff 2 to 3 weeks after the invitation to encourage screening completion.
  Centralized processes to promote guideline-based follow-up.
  Arms: FIT Screening Strategy
Other: Choice Screening Strategy — Mailed outreach invitation offering patients the choice to complete either a FIT or schedule a colonoscopy.
  Letter will discuss advantages and disadvantages of FIT vs. colonoscopy but will not recommend a particular test, allowing patients to choose a screening option based on their own preferences. Outreach includes: 1) invitation letter, 2) choice grid 3) telephone number for scheduling colonoscopy, and 4) test kit (1-sample FIT, simplified instructions on how to perform the test and return mailer with prepaid postage).
  Up to three "live" phone call reminders from project staff 2 to 3 weeks after the mailed invitation to encourage screening completion.
  Centralized processes to promote guideline-based follow-up.
  Arms: Choice Screening Strategy

SUMMARY:
This is a pragmatic, randomized, controlled trial comparing whether a mailed outreach intervention offering patients who are not up-to-date with colorectal cancer (CRC) a choice of completing a home Fecal Immunochemical Test (FIT) test or scheduling a screening colonoscopy increases CRC screening completion compared to a mailed FIT kit outreach program (which does not offer an explicit choice of screening modality). The trial will be conducted in a racially and socioeconomically diverse cohort of patients served by an integrated safety net delivery system that has a "FIT first" population health screening strategy. All patients will also have access to whatever CRC screening is recommended through usual visit-based care.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the 2nd leading cause of cancer death in the US, though CRC death can be reduced by screening. In the NCI-funded UT Southwestern-Parkland PROSPR Center (U54 CA163308), mailed FIT-based outreach doubled the proportion of patients up-to-date with screening compared to usual care. Investigators are now conducting a comparative effectiveness trial to evaluate the effect of a mailed invite offering a choice of FIT or colonoscopy (n=2,000) on one-time CRC screening completion compared to mailed FIT-based outreach (which does not offer an explicit choice of screening modality (n=8,000.) Randomization will be stratified based on whether or not patients completed a FIT within the prior 18-month period. Patients randomized to FIT outreach will receive: a) low-literacy educational letters, b) mailed screening outreach invitations, c) a one-sample home FIT kit and return mailer with prepaid postage, d) telephone reminder calls including one-on-one education, and e) centralized patient navigation for follow-up of abnormal screening results, and treatment for patients newly diagnosed with CRC. Patients randomized to the "choice" arm will receive the same materials described above; however, the educational letter will explain and offer the additional choice of screening by colonoscopy (instead of completing the mailed FIT kit). The mailing will include a low health literacy one-page option grid outlining the pros and cons of FIT vs. colonoscopy. We will not recommend a particular test as preferred but instead emphasize that both are good choices, and the patient should choose the screening option that seems right for them. Patients choosing colonoscopy will be provided a telephone number to schedule the procedure. During scheduling, patients will be triaged by study staff with a structured history and physical form to "direct access" colonoscopy or a pre-colonoscopy clinic visit. Patients choosing FIT can return the one-sample mailed FIT kit using the return envelope with prepaid postage.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Age 50-64 years
* Seen at least one time at a Parkland primary care clinic within one year prior to randomization
* Participants in Parkland's medical assistance program for the uninsured (Parkland Financial Assistance)
* All races and ethnicities

Exclusion Criteria:

* Up-to-date with CRC screening, defined by:

  1. Colonoscopy in the last 10 years
  2. Sigmoidoscopy in the last 5 years
* Prior history of CRC, total colectomy, inflammatory bowel disease, or colon polyps
* Address or phone number not on file
* Incarcerated

Ages: 50 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26859 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
One-time Screening Completion | Within one year of randomization
  Proportion of patients who complete CRC screening with colonoscopy, sigmoidoscopy, or FIT

SECONDARY OUTCOMES:
Screening Up-to-date | At 2 and 3 years post-randomization
  Screening Up-to-date status
Choice of FIT versus Colonoscopy | Within 6 months of invitation
  Proportion of patients who choose FIT versus colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Amit Singal, MD, MS, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Health & Hospital System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No